CLINICAL TRIAL: NCT03080155
Title: Evaluation of a Three Dimensional Functional Metabolic Imaging and Risk Assessment System in Classifying Women for Likelihood of Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Real Imaging Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 960-CLP-GER_Multimodality_GER1
Record Dates: First submitted 2017-03-07; First posted 2017-03-15 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIRA device imaging (Experimental): MIRA Device imaging for adjunctive detection of breast cancer
  Interventions: Device: MIRA device imaging

INTERVENTIONS:
Device: MIRA device imaging — MIRA Device imaging for adjunctive detection of breast cancer
  Other Names: Real Imager 8

SUMMARY:
The purpose of the study is to assess the effectiveness of MIRA in classifying women with dense breast tissue for supplemental breast MRI. To assess the effectiveness of MIRA for correctly classifying women with breast cancer and to evaluate the safety of the device.

In women above 30 years old who are undergoing MRI or are scheduled for image-guided needle biopsy due to lesions detected by other imaging modalities.

ELIGIBILITY:
Inclusion Criteria:

* Women who are between 30 to 70 years of age and who are asymptomatic and scheduled to undergo routine breast cancer screening (MRI and/or mammography) OR
* Women who are between 30 to 79 years of age and scheduled for image-guided needle biopsy as a result of findings obtained during standard of care imaging modalities (mammography, ultrasound and/or MRI) performed at the clinical site that participates in the study.

Exclusion Criteria:

1. Contraindication to bilateral mammography or MRI.
2. Subjects who are unable to read, understand and execute the informed consent procedure.
3. Subjects who have had mammography, ultrasound or MRI examination performed on the day of the study prior to MIRA scan.
4. Subjects who have significant existing breast trauma.
5. Subjects who have undergone lumpectomy/mastectomy.
6. Subjects who have undergone breast reduction or breast augmentation.
7. Subjects who have undergone any other type of breast surgery.
8. Subjects who have large breast scar / Breast deformation.
9. Subjects who have undergone a breast needle biopsy within the 6-month period prior to their intended enrollment into the study.
10. Subjects who have a temperature > 37.8C degrees on the day of the MIRA imaging.
11. Subjects who are pregnant or lactating.
12. Subjects who have had placement of an internal breast marker.
13. Subjects with known Raynaud's Disease.
14. Subjects that are claustrophobic or have physical limitations that do not allow them to sit in the system chair for the required imaging session.
15. Subjects with implanted pacemaker/defibrillator, implanted venous access device (portacath) or other implanted devices.
16. Inmates or mentally disabled individuals.
17. Subjects with a BI-RADS category 6 (e.g. for which mammogram was performed for the purpose of planning cancer therapy).
18. Subjects who participated in the Calibration Phase will not be able to participate in the Testing Phase.
19. Subjects currently participating in another investigational clinical study.
20. Subjects undergoing breast MR for pre-staging.
21. Subjects with known Mastitis

Ages: 30 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
determining MIRA's PPV (positive predictive value) | 24 months
  * The positive predictive value (and the amount of false-positive diagnoses) of MIRA will be determined using positive MRI (MRI BI-RADS >= 3) as a reference test in cohort of women with negative (Mammography BI-RADS 1 or 2).
  * The positive predictive value (and the amount of false-positive diagnoses) of MIRA will be determined using the histological diagnosis as the reference test in ALL women participated in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Fischer, Prof., Principal Investigator — BrustZentrum, Göttingen
Locations (1):
- BrustZentrum, Göttingen, Germany